CLINICAL TRIAL: NCT05546866
Title: An Open-label, Prospective, Multi-center, Single-arm Study to Assess the Efficacy and Safety of Adjuvant Osimertinib in Non-small Cell Lung Cancer (NSCLC) With Uncommon Epidermal Growth Factor Receptor Mutations (EGFRm)
Brief Title: Study to Assess the Efficacy and Safety of Adjuvant Osimertinib in NSCLC With Uncommon EGFRm
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5161C00024
Record Dates: First submitted 2022-03-11; First posted 2022-09-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osimertinib (Experimental): Subjects successfully enrolled into the study will receive 80mg osimertinib QD p.o. until completion of planned treatment duration, recurrence of disease, or other treatment discontinuation criteria is met. The maximum treatment duration period is 3 years.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Subjects successfully enrolled into the study will receive 80mg osimertinib QD p.o. until completion of planned treatment duration, recurrence of disease, or other treatment discontinuation criteria is met. The maximum treatment duration period is 3 years.

SUMMARY:
This is an open-label, multi-centre, single-arm study assessing the efficacy and safety of osimertinib as adjuvant treatment in stage IB-IIIB (8th AJCC) NSCLC with uncommon EGFRm after receiving complete surgical resection with or without adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures, sampling, and analyses.
2. Male or female, aged at least 18 years.
3. Histologically confirmed diagnosis of primary non-small cell lung cancer (NSCLC) on predominantly non-squamous histology.
4. MRI or CT scan of the brain must be done prior to surgery as it is considered standard of care. Patients in whom this was not done prior to surgery may still be enrolled if appropriate imaging is performed prior to enrollment.
5. Patients must be classified post-operatively as Stage IB, II, IIIA, or IIIB on the basis of pathologic criteria. Staging will be according to the 8th edition of AJCC Cancer Staging Manual.
6. At least one documented uncommon EGFR mutation of G719X/L861Q/S768I/de novo T790M without EGFR Ex19del/L858R/exon 20 insertion as detected in tumour tissue, through real-time PCR or NGS analysis from accredited laboratories approved by the Chinese regulatory authority.
7. Complete surgical resection of the primary NSCLC is mandatory. All gross disease must have been removed at the end of surgery. All surgical margins of resection must be negative for tumour. Resection may be accomplished by open or Video Associated Thoracic Surgery (VATS) techniques.
8. Complete recovery from surgery and standard post-operative therapy (if applicable) at the time of enrollment. Treatment cannot commence within 4 weeks following surgery. No more than 10 weeks may have elapsed between surgery and the enrollment for patients who have not received adjuvant chemotherapy; no more than 26 weeks may have elapsed between surgery and enrollment for patients who received adjuvant chemotherapy.

   * Complete post-operative wound healing must have occurred following any surgery.
   * For patients who received post-operative adjuvant platinum-based chemotherapy, a minimum of 2 weeks must have elapsed (but no more than 10 weeks) from the last administered dose of chemotherapy to the date of enrollment.
   * Patients must have recovered from all toxicities of prior therapy greater than CTCAE Grade 1 at the time of starting study treatment with the exception of alopecia and Grade 2 prior platinum therapy related neuropathy.
9. World Health Organization Performance Status of 0 to 1.
10. Females must be using highly effective contraceptive measures, and must have a negative pregnancy test prior to start of dosing if of child-bearing potential, or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

    * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
    * Women less than 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the institution.
    * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation.

    Further information in Appendix D (Definition of Women of Childbearing Potential and Acceptable Contraceptive Methods) Male patients must be willing to use barrier contraception, (see Restrictions, Section 5.3).
11. For inclusion in the optional part in molecular research study, patients must provide informed consent for the optional analysis.

If a patient declines to participate in any voluntary exploratory research of the study, there will be no penalty or loss of benefit to the patient and he/she will not be excluded from other aspects of the study.

Exclusion Criteria:

1. Previous enrollment and treatment in the present study.
2. Participation in another clinical study with a study intervention or investigational medicinal device administered in the last 8 weeks prior to enrollment, or concurrent enrollment and exposure in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
3. Treatment with any of the following:

   * Pre-operative or post-operative or planned radiation therapy for the current lung cancer.
   * Pre-operative (neo-adjuvant) platinum based or other chemotherapy.
   * Any prior anticancer therapy, including investigational therapy, for treatment of NSCLC other than standard platinum based doublet post-operative adjuvant chemotherapy.
   * Prior treatment with neoadjuvant or adjuvant EGFR-TKI.
   * Major surgery (including primary tumour surgery, excluding placement of vascular access) within 4 weeks of the first dose of study drug.
   * Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inducers of CYP3A4 (at least 3 week prior) (Appendix F). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4.
   * Treatment with an investigational drug within five half-lives of the compound or any of its related material, if known.
4. Patients who have had only segmentectomies or wedge resections.
5. History of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer, or other solid tumours curatively treated with no evidence of disease for > 5 years following the end of treatment and which, in the opinion of the treating physician, do not have a substantial risk of recurrence of the prior malignancy.
6. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol; or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).

   * Screening for chronic conditions is not required.
   * Active infection will include any patients receiving treatment for infection.
   * Subjects with a resolved or chronic infection HBV are eligible if they are:

     1. Negative for HBsAg and positive for hepatitis B core antibody [anti-HBc IgG] or
     2. Positive for HBsAg, negative for HBeAg but for > 6 months have had transaminases levels below ULN and HBV DNA levels ≤ 100 IU/mL (i.e., are in an inactive carrier state). Refer to Restrictions, Section 5.3.
7. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of osimertinib.
8. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) >470 msec, obtained from 3 ECGs, using the screening clinic ECG machine-derived QTcF value.
   * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG, e.g., complete left bundle branch block, third-degree heart block, second-degree heart block.
   * Patient with any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as electrolyte abnormalities* including:
   * Serum/plasma potassium < LLN
   * Serum/plasma magnesium < LLN
   * Serum/plasma calcium < LLN heart failure, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsades de Pointes (TdP) .

     * Note: Correction of electrolyte abnormalities to within normal ranges can be performed during the screening period.
9. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
10. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

    * Absolute neutrophil count <1.5 × 109/L.
    * Platelet count <100 × 109/L.
    * Haemoglobin <90 g/L.
    * Alanine aminotransferase (ALT) >2.5× the upper limit of normal (ULN).
    * Aspartate aminotransferase (AST) >2.5 × ULN.
    * Total bilirubin >1.5 × ULN or >3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia).
    * Creatinine >1.5 × ULN concurrent with creatinine clearance <50 mL/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 × ULN.
11. History of hypersensitivity to active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib.
12. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
13. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca representative and/or staff at the study site).
14. Currently pregnant (confirmed with positive pregnancy test) or breast feeding.

In addition, the following are considered criteria for exclusion from the exploratory molecular research only:

1. Prior allogeneic bone marrow transplant.
2. Non-leukocyte depleted whole blood transfusion within 120 days of sample collection.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival (DFS) rate by investigator assessment | Up to 3 years for each subject from the first dosing of study treatment.
  DFS is defined as the time from the first dosing of study treatment until the date of disease recurrence by investigator assessment or death by any cause in the absence of disease recurrence. DFS rate at 3 years is defined as the proportion of patients alive and disease free at 3 years from the first dosing of study treatment as estimated by Kaplan-Meier method, respectively. Patients who are disease-free and alive at the time of analysis will be censored at the date of their latest follow-up assessment known to be disease-free

SECONDARY OUTCOMES:
DFS rate at 2 years | Up to 2 years for each subject from the first dosing of study treatment.
  DFS is defined as the time from the first dosing of study treatment until the date of disease recurrence by investigator assessment or death by any cause in the absence of disease recurrence. DFS rate at 2 years is defined as the proportion of patients alive and disease free at 2 years from the first dosing of study treatment as estimated by Kaplan-Meier method, respectively. Patients who are disease-free and alive at the time of analysis will be censored at the date of their latest follow-up assessment known to be disease-free.
DFS rate at 5 years | Up to 5 years for each subject from the first dosing of study treatment.
  DFS is defined as the time from the first dosing of study treatment until the date of disease recurrence by investigator assessment or death by any cause in the absence of disease recurrence. DFS rate at 5 years is defined as the proportion of patients alive and disease free at 5 years from the first dosing of study treatment as estimated by Kaplan-Meier method, respectively. Patients who are disease-free and alive at the time of analysis will be censored at the date of their latest follow-up assessment known to be disease-free.
OS rate at 2 years | Up to 2 years for each subject from the first dosing of study treatment.
  OS (Overall survival) is defined as the time from the first dosing of study treatment to the date of death from any cause; OS rate at 2 years is defined as the proportion of patients alive at 2 years from the first dosing of study treatment; Following disease recurrence, patients will be followed up for survival every 24 weeks until study completion
OS rate at 3 years | Up to 3 years for each subject from the first dosing of study treatment.
  OS (Overall survival) is defined as the time from the first dosing of study treatment to the date of death from any cause; OS rate at 3 years is defined as the proportion of patients alive at 3 years from the first dosing of study treatment; Following disease recurrence, patients will be followed up for survival every 24 weeks until study completion
OS rate at 4 years | Up to 4 years for each subject from the first dosing of study treatment.
  OS (Overall survival) is defined as the time from the first dosing of study treatment to the date of death from any cause; OS rate at 4 years is defined as the proportion of patients alive at 4 years from the first dosing of study treatment; Following disease recurrence, patients will be followed up for survival every 24 weeks until study completion
OS rate at 5 years | Up to 5 years for each subject from the first dosing of study treatment.
  OS (Overall survival) is defined as the time from the first dosing of study treatment to the date of death from any cause; OS rate at 5 years is defined as the proportion of patients alive at 5 years from the first dosing of study treatment; Following disease recurrence, patients will be followed up for survival every 24 weeks until study completion
Median DFS by investigator assessment (if applicable) | Up to 5 years for each subject from the first dosing of study treatment.
  DFS is defined as the date from first dosing of study treatment until the date of disease recurrence by investigator assessment or death from any cause in the absence of disease recurrence.Patients will be evaluated for disease recurrence at 12 weeks, 24 weeks, relative to enrollment, and then every 24 weeks until recurrence or 5 years. It is important to follow the assessment schedule as closely as possible.
DFS rate at 4 years | Up to 4 years for each subject from the first dosing of study treatment.
  DFS is defined as the time from the first dosing of study treatment until the date of disease recurrence by investigator assessment or death by any cause in the absence of disease recurrence. DFS rate at 4 years is defined as the proportion of patients alive and disease free at 4 years from the first dosing of study treatment as estimated by Kaplan-Meier method, respectively. Patients who are disease-free and alive at the time of analysis will be censored at the date of their latest follow-up assessment known to be disease-free.

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Kunming
  - Research Site, Ningbo
  - Research Site, Shijiazhuang
  - Research Site, Suzhou
  - Research Site, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home